CLINICAL TRIAL: NCT06514430
Title: Prophylactic Analgesia in Outpatient Intradetrusor onabotulinumtoxinA Injections: Efficacy and Feasibility of Alternative Pain Control Methods in a Diverse Urban Patient Population
Brief Title: Prophylactic Analgesia for Bladder Botox Injections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: It was determined that it would be impracticable to conduct this study as a randomized trial. Study has been repurposed as a non-randomized study.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-16001
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Urge; Overactive Bladder
Keywords: onabotulinumtoxinA (Botox) injection; oral phenazopyridine; intravesical lidocaine; Urban Patient Population; Analgesia; Pain Management; Diverse Populations
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge; Urinary Bladder, Overactive; Agnosia | interventions — Phenazopyridine; Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral phenazopyridine (Active Comparator): Patients randomized to the oral phenzopyridine arm will receive 200 milligrams (mg) phenazopyridine orally prior to the scheduled procedure.
  Interventions: Drug: Phenazopyridine
- Intravesical lidocaine (Active Comparator): Patients randomized to the intravesical lidocaine arm will be administered 50 cubic centimeters (cc) of 1% lidocaine with 50cc sodium bicarbonate within the bladder immediately prior to the procedure.
  Interventions: Drug: 1% lidocaine with sodium bicarbonate

INTERVENTIONS:
Drug: Phenazopyridine — 200mg PO Phenazopyridine taken prior to the Botox® injection procedure as an analgesic.
  Other Names: Pyridium
  Arms: Oral phenazopyridine
Drug: 1% lidocaine with sodium bicarbonate — 50cc of 1% lidocaine with 50cc sodium bicarbonate injected into the bladder lumen prior to the Botox® injection procedure.
  Other Names: Intravesical lidocaine
  Arms: Intravesical lidocaine

SUMMARY:
The goal of this clinical trial is to learn more about using phenazopyridine (Pyridium) for pain control during bladder onabotulinumtoxinA ("botox") injections for surgical management of overactive bladder (OAB) for patients at Montefiore Medical Center in The Bronx. It will also learn about if using the phenazopyridine pill affects how satisfied patients are with their experience, how much pain patients feel afterwards, and if doctors think using the Pyridium pill affected how they performed the procedure. The main question it aims to answer is:

- Is oral phenazopyridine at least as good as intravesical lidocaine is for managing pain with bladder botox injections for OAB in Montefiore patients?

Researchers will compare phenazopyridine to intravesical lidocaine, a liquid put into the bladder, to see if phenazopyridine is at least as good at controlling pain with bladder botox injections as intravesical lidocaine is.

Participants will be assigned, by chance, to receive either the oral phenazopyridine pill or the intravesical lidocaine as their pain control for the procedure.

DETAILED DESCRIPTION:
Urinary incontinence poses personal and emotional hardships to the patients who experience it. Urge urinary incontinence (UUI) is often a result of overactive bladder (OAB) and may exist in combination with stress urinary incontinence (SUI), termed mixed urinary incontinence (MUI). Overall, it is estimated that 25-45% of women experience some degree of urinary incontinence (UI), with increasing prevalence of UI symptoms as women age. Treatment options for UI include expectant management, behavioral modification, pelvic floor physical therapy, continence pessary, vaginal inserts, colposuspension or sling insertion, as well as intradetrusor onabotulinumtoxinA ("botox") injections and urethral bulking procedures.

While intradetrusor onabotulinumtoxinA injection is a viable and effective option for OAB, little is known about effective pain management for patients undergoing this procedure. To date, there has not yet been research on analgesia for bladder Botox injections in diverse, urban populations whose needs and experience of pain may differ from those of other patients. In recent years, there has been renewed attention among patients and discussion within medical communities on the importance of examining biological sex, gender, racial, and ethnic disparities in acute pain management.

In this randomized controlled trial (RCT), the use of oral phenazopyridine compared to intravesical lidocaine as analgesic options for Montefiore patients undergoing surgical management of idiopathic overactive bladder with intradetrusor onabotulinumtoxinA (Botox) injections at the Department of Female Pelvic Medicine and Reconstructive Surgery in the Bronx, will be studied. Oral phenazopyridine is a pre-1938 FDA grandfathered drug that will be utilized in accordance with its indication for the treatment of urinary pain in the outpatient setting. The use of these less invasive but effective analgesic options to manage pain for outpatient urogynecological procedures and their acceptability in a diverse, urban patient population will be examined.

All pain control options included in this study are within the standard of care for bladder Botox injections. Participants will not have any alteration in their clinical care from what would be experienced if not participating in the study other than being randomized to one analgesia protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years or older
* Planning to undergo surgical management of idiopathic overactive bladder with intradetrusor onabotulinumtoxinA injection at Montefiore Medical Center Female Pelvic Medicine Reconstructive Surgery Department
* Provided informed consent

Exclusion Criteria:

* Currently pregnant
* Current Urinary Tract Infection (UTI)
* Neurogenic bladder diagnosis
* Received pelvic radiotherapy
* Severe cognitive impairment
* Non-English or non-Spanish speaking.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Bladder Pain | Day of the procedure
  Patient-reported bladder pain will be assessed using the Visual Analog Quality of Life Scale (VAS) tool. The VAS is a unidimensional measure of pain intensity. The 100mm VAS intervention tool consists of an emoji face scale ranging from an "open-mouth smile" emoji to a crying emoji. Patients will place an 'x' on the number line below the emojis to indicate where on the scale they would rate their pain, using the emoji faces as a guide. The distance from the lowest (farthest left) point on this scale to the 'x' will be measured and reported in millimeters. Higher scores are associated with increased levels of bladder pain intensity. Group median pain scores will be tabulated and reported.

SECONDARY OUTCOMES:
Patient satisfaction | 3 days post-procedure
  Overall patient satisfaction will be measured using a 5-point Likert scale range where 5 = very satisfied; 4 = satisfied; 3= neutral; 2 = unsatisfied; and 1 = very unsatisfied. Overall group mean patient satisfaction scores will be summarized and reported. Higher scores are associated with increased levels of patient satisfaction.
Bladder visualization | Day of the procedure
  Physicians will be queried as to their perception of bladder visualization following the procedure, as oral phenazopyridine is known to temporarily stain the urine orange. Bladder visualization will be performed using cystoscopy to view the inside of the bladder during the procedure. Bladder visualization will be assessed on the following scale: 0 = clear, no difficulty; 1 = somewhat difficult / mildly impaired, 2 = very difficult.
Bladder Pain | 3 days post-operation
  Patient-reported bladder pain will be assessed using the Visual Analog Quality of Life Scale (VAS) tool. The VAS is a unidimensional measure of pain intensity. The 100mm VAS intervention tool consists of an emoji face scale ranging from an "open-mouth smile" emoji to a crying emoji. Patients will place an 'x' on the number line below the emojis to indicate where on the scale they would rate their pain, using the emoji faces as a guide. The distance from the lowest (farthest left) point on this scale to the 'x' will be measured and reported in millimeters. Higher scores are associated with increased levels of bladder pain intensity. Group median pain scores will be tabulated and reported.
Postoperative Analgesia | 3 days post-operation
  Self-reported use of additional analgesia immediately following the procedure will be evaluated as 0 = no additional analgesia and 1 = any additional analgesia. The number of patients who require any additional postoperative analgesic will be summarized and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Laudano, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center Female Pelvic Medicine Reconstructive Surgery Department, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No